CLINICAL TRIAL: NCT05148858
Title: Study the Patterns of Sleep Disturbance and Quality of Life During Corona Virus Disease 19 (COVID 19) Pandemic in Upper Egypt
Brief Title: Sleep Quality and Quality of Life in Coronavirus 19 Disease ( COVID 19) Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Manal Mahmoud, Principal Investigator, Assiut University
Other Study IDs: Qol in Covid
Record Dates: First submitted 2021-11-16; First posted 2021-12-08 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2021-12

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases: Patients affected by COVID-19 infection
- Control: Normal subjects not affected by COVID-19 infection

SUMMARY:
To study the impact of COVID 19 infection on sleep habit as regards quality of sleep, emergence of insomnia.

To assess quality of life in patients after COVID 19 infection.

DETAILED DESCRIPTION:
The year 2020 will be remembered for a cataclysmic event- the coronavirus disease 19 ( COVID 19) pandemic, caused by severe acute respiratory syndrome coronavirus 2.

COVID 19 is a serious disease that can significantly affect the daily lives of recovered patients and their families in terms of mental health problems such as post- traumatic stress, depression, anxiety, and insomnia, as well as the negative impact COVID 19 has on patients quality of life. Since the patients are not immune to future infection, it may lead to a more negative impact on patient's quality of life. Health related quality of life is an important measure that is used for assessing the impact of diseases, disorders, or disabilities on the physical, mental, and social domains of patients health. The assessment of health related quality of life (HRQol) helps healthcare providers identify the factors affecting quality of life (QoL) and recognize the aspects of COVID 19 management that needs to be enhanced for improving the QoL of patients. COVID 19 infection causes systemic inflammation leading to a surge on inflammatory mediators in the body that are known to influence sleep and vice versa.

Systemic infection related increase in the inflammatory mediators are known to increase the amount of non rapid eye movement (NREM) sleep and duration of sleep, perhaps in an attempt to save energy and counter the infection. However, different infections have varying effects on sleep. That could be one reason that COVID 19 infection has led to insomnia and worsening of sleep quality rather than increment in sleep. Not only the sleep quality has been affected during the COVID 19 pandemic, but pandemic could have led to emergence of sleep disorders as well.

It has been persuasively argued as to why elderly persons are more susceptible to contract severe acute respiratory syndrome coronavirus 2 (SARS-COV-2) infection. Several factors have been discussed that worsens sleep among the elderly, including aging of the circadian network.

Considering high prevalence of these disorders, optimal management of these disorders is important during pandemic not only to reduce the risk of contracting SARS-COV-2 infection, but also to reduce adverse health consequences related to same.

This is an important area for research as the relationship appears bidirectional, improvement in sleep may be used to reduce impact of COVID 19 and vice versa.

ELIGIBILITY:
Inclusion Criteria:

* Mild, moderate and severe COVID 19 cases will be included in our study. Either diagnosed by polymerase chain reaction (PCR), CT changes characteristic of COVID 19 infection or by symptomatology and laboratory investigations.

Either managed as an outpatient or admitted to hospital. Either admitted to ward or to ICU. Age above 18 years old. With no history of end stage organ failure. With no history of neurological, psychiatric disease or cerebrovascular insufficiency.

Exclusion Criteria:

* Age below 18 years old. End stage organ failure. Patients with neurological, psychiatric diseases and cerebrovascular insufficiency.

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mild, moderate and severe COVID 19 cases above 18 years old with no history of neurological, psychiatric disease or cerebrovascular insufficiency with no history of end stage organ failure.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-04-01 (Estimated); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Quality of life in coronavirus 19 disease ( COVID-19) patients | One month after the infection
  Euro quality of life (Euro QoL) questionnaire in which higher scores mean a worse outcome.
  Minimum value is 11111 Maximum value is 55555

SECONDARY OUTCOMES:
To assess quality of sleep in coronavirus 19 ( COVID-19) patients using Epworth sleepiness scale (ESS). | One month after infection
  ESS in which higher scores mean worse outcomes. ESS minimum value is zero, while maximum value is 24
To assess quality of sleep in coronavirus 19 ( COVID-19) patients using Pittsburgh sleep quality index ( PSQI) | One month after the infection.
  PSQI in which higher scores mean worse outcomes. PSQI minimum value is zero, while maximum value is 21

CONTACTS AND LOCATIONS:
Overall Officials: Manal Mahmoud, Principal Investigator — Assiut University

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, Ho CS, Ho RC. Immediate Psychological Responses and Associated Factors during the Initial Stage of the 2019 Coronavirus Disease (COVID-19) Epidemic among the General Population in China. Int J Environ Res Public Health. 2020 Mar 6;17(5):1729. doi: 10.3390/ijerph17051729. PMID 32155789
- [Background] Wang C, Pan R, Wan X, Tan Y, Xu L, McIntyre RS, Choo FN, Tran B, Ho R, Sharma VK, Ho C. A longitudinal study on the mental health of general population during the COVID-19 epidemic in China. Brain Behav Immun. 2020 Jul;87:40-48. doi: 10.1016/j.bbi.2020.04.028. Epub 2020 Apr 13. PMID 32298802
- [Background] Tan BYQ, Chew NWS, Lee GKH, Jing M, Goh Y, Yeo LLL, Zhang K, Chin HK, Ahmad A, Khan FA, Shanmugam GN, Chan BPL, Sunny S, Chandra B, Ong JJY, Paliwal PR, Wong LYH, Sagayanathan R, Chen JT, Ng AYY, Teoh HL, Ho CS, Ho RC, Sharma VK. Psychological Impact of the COVID-19 Pandemic on Health Care Workers in Singapore. Ann Intern Med. 2020 Aug 18;173(4):317-320. doi: 10.7326/M20-1083. Epub 2020 Apr 6. No abstract available. PMID 32251513
- [Background] Hao F, Tan W, Jiang L, Zhang L, Zhao X, Zou Y, Hu Y, Luo X, Jiang X, McIntyre RS, Tran B, Sun J, Zhang Z, Ho R, Ho C, Tam W. Do psychiatric patients experience more psychiatric symptoms during COVID-19 pandemic and lockdown? A case-control study with service and research implications for immunopsychiatry. Brain Behav Immun. 2020 Jul;87:100-106. doi: 10.1016/j.bbi.2020.04.069. Epub 2020 Apr 27. PMID 32353518
- [Background] Nguyen HC, Nguyen MH, Do BN, Tran CQ, Nguyen TTP, Pham KM, Pham LV, Tran KV, Duong TT, Tran TV, Duong TH, Nguyen TT, Nguyen QH, Hoang TM, Nguyen KT, Pham TTM, Yang SH, Chao JC, Duong TV. People with Suspected COVID-19 Symptoms Were More Likely Depressed and Had Lower Health-Related Quality of Life: The Potential Benefit of Health Literacy. J Clin Med. 2020 Mar 31;9(4):965. doi: 10.3390/jcm9040965. PMID 32244415
- [Background] Ameri H, Yousefi M, Yaseri M, Nahvijou A, Arab M, Akbari Sari A. Mapping the cancer-specific QLQ-C30 onto the generic EQ-5D-5L and SF-6D in colorectal cancer patients. Expert Rev Pharmacoecon Outcomes Res. 2019 Feb;19(1):89-96. doi: 10.1080/14737167.2018.1517046. Epub 2018 Sep 3. PMID 30173585
- [Background] Ibarra-Coronado EG, Pantaleon-Martinez AM, Velazquez-Moctezuma J, Prospero-Garcia O, Mendez-Diaz M, Perez-Tapia M, Pavon L, Morales-Montor J. The Bidirectional Relationship between Sleep and Immunity against Infections. J Immunol Res. 2015;2015:678164. doi: 10.1155/2015/678164. Epub 2015 Aug 31. PMID 26417606
- [Background] Cardinali DP, Brown GM, Reiter RJ, Pandi-Perumal SR. Elderly as a High-risk Group during COVID-19 Pandemic: Effect of Circadian Misalignment, Sleep Dysregulation and Melatonin Administration. Sleep Vigil. 2020;4(2):81-87. doi: 10.1007/s41782-020-00111-7. Epub 2020 Sep 26. PMID 33015537
- [Background] Shrivastava D. Unprecedented Events do not Always Call for Unprecedented Actions. Sleep Vigil. 2020;4(1):1-2. doi: 10.1007/s41782-020-00088-3. Epub 2020 May 25. No abstract available. PMID 32838114
- [Background] Sullivan CE. Snoring and obstructive sleep apnoea as risk factors in SARS-Cov-2: can nasal CPAP during sleep reduce pneumonia risk? Sleep Biol Rhythms. 2021;19(1):109-110. doi: 10.1007/s41105-020-00295-5. Epub 2020 Nov 7. No abstract available. PMID 33192172